CLINICAL TRIAL: NCT06025058
Title: Researcher-led Clinical Study to Evaluate the Effectiveness and Safety of the Application of Neopep-S-based Easy Dew MD Regen Cream in Patients Under Radiotherapy After Breast Tumor Resection
Brief Title: Neopep-S-based EasyDew MD Regen Cream for Radiotherapy Subject After Breast Tumor Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eun-ji Kim (Industry)
Responsible Party: Sponsor-Investigator, Eun-ji Kim, Clinical Trial Manager, CGBio Inc.
Organization: CGBio Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: G2207
Record Dates: First submitted 2023-08-25; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Skin Lesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Easy Dew MD Regen Cream (Experimental): In the case of the study group among the subjects of the clinical study, The experimental group apply an appropriate amount of EasyDew MD Regen Cream twice a day (morning and evening) and can be absorbed well.
  Interventions: Device: Easy Dew MD Regen Cream
- Physiogel Stability Intensive Cream MD (Active Comparator): The subject applies the provided medical device twice a day (morning and evening) to areas with symptoms of dry skin so that it can be absorbed well.
  Interventions: Device: Easy Dew MD Regen Cream

INTERVENTIONS:
Device: Easy Dew MD Regen Cream — The subject applies the provided medical device twice a day (morning and evening) to areas with symptoms of dry skin so that it can be absorbed well.
  Other Names: Physiogel Stability Intensive Cream MD

SUMMARY:
This clinical study is conducted prospectively for 3 months after medical device treatment. It is a comparative clinical study of the leading control group.

DETAILED DESCRIPTION:
Subject is a patient who has a tumor removed from the breast and is receiving radiotherapy at the lesion.

Subjects (and/or legal representatives) have agreed in writing to participate in the clinical study.

Perform a post-screening test. Evaluating the screening test results, meeting the selection criteria, and meeting the exclusion criteria.

Those who do not are registered for clinical research.

* Control group: Physiogel Skin Stability Intensive Cream MD (10 people)
* Study Group: EasyDew MD Regen Cream (20 people) The subjects of the clinical study are randomly assigned in a 2:1 ratio between the study group and the control group.

In this case, apply the control medical device twice a day (morning and evening) to the radiation treatment area.

Apply it. In the case of the research group, easy dew MD Regen Cream was applied to the radiotherapy site.

Apply an appropriate amount twice a day (in the evening) to ensure good absorption.

The progress for three months after the application of medical devices for clinical research will be observed, and the subjects will be screening visit (Visit1), medical device application day (Visit2), medical device application, and medical device application.

Visit the research institution regularly for one month (Visit3) and three months after application (Visit4) for validity and to be evaluated for safety.

ELIGIBILITY:
Inclusion Criteria:

* adults over the age of 19
* The tumor in the breast area is resected and radiotherapy is planned, performed, or Subjects with a history of irradiation
* Decide to participate in this clinical study arbitrarily and in the written informed consent a person to whom

Exclusion Criteria:

* When participating in a clinical study, the findings of radiation dermatitis in the area are shown
* A person who shows signs of acute or chronic dermatological diseases
* In situations where the requirements of a clinical study cannot be complied with
* When the researcher's judgment determines that the participation of the study is inappropriate (e.g. Kelloid personality)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Transepidermal water loss | before and one month, 3month after medical device application with GP SKin(machine/measuring the degree of moisture skin water loss)
  Percutaneous moisture loss measured

SECONDARY OUTCOMES:
Itching score | Before, after one month after application, 3 month after application
  Evaluate the Itching scale / lowest 1 score ( best score) to highest 5 score( worst
VSS | Before, after one month after application, 3 month after application
  Vancouver Scar Scale/ No range of upper and lower score, the lower is best
BREAST-Q Survey Assessment | Before, after one month after application, 3 month after application
  Evaluate the BREAST-Q Survey Assessment/ lowest 1 score (worst) to highest 10 score( best score)

CONTACTS AND LOCATIONS:
Overall Officials: Jihye Lee, Master, Study Director — CGBio Inc.
Locations (1):
- Ajou University Hospital, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No